CLINICAL TRIAL: NCT05997472
Title: The Effect of The Use of Walking Aid On Timed Up and Go Test In Patients With Stroke
Brief Title: The Effect of Using Walking Aid On TUG Test
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Esra KESKİN, Research Assisstant, Bandırma Onyedi Eylül University
Other Study IDs: 2023-122
Record Dates: First submitted 2023-08-08; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Locomotion Disorder, Neurologic
Keywords: stroke; Timed Up and Go Test; balance; locomotion
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: evaluation af mobility and balance — evaluation af mobility and balance Timed Up and Go Test Berg Balance Scale

SUMMARY:
The Timed Up and Go Test is a measurement tool that allows the participant to use assistive devices and walking aids during the test that evaluates functional mobility. This study was conducted to determine the effect of using walking aids on the Timed Up and Go test and it's correlation with balance in stroke patients.

DETAILED DESCRIPTION:
Cross-sectional, observational study

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Test >24
* Stroke patients who can walk 10 meters with or without walking aid

Exclusion Criteria:

* Individuals dependent on bed or wheelchair
* Individuals with musculoskeletal disease that may adversely affect mobility and balance.
* Individuals who have had any operation in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients older than 18 years of age at least 6 weeks after stroke
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-08-21 (Estimated); Study Completion 2023-10-21 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test | up to 4 weeks
  Mobility

SECONDARY OUTCOMES:
Berg Balance Scale | up to 4 weeks
  Balance

CONTACTS AND LOCATIONS:
Overall Officials: EBRU KAYA MUTLU, Study Chair — BANDIRMA ONYEDİ EYLÜL UNIVERSITY
Locations (1):
- Bandirma Onyedi Eylül University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No